CLINICAL TRIAL: NCT01476046
Title: A Two-part, Randomised, Placebo-controlled Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamicsof Single and Repeat Doses of Intravenously Infused GSK1995057 in Healthy Subjects.
Brief Title: Safety Study of GSK1995057 Given as Single and Repeat Intravenous Doses in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 110951
Record Dates: First submitted 2011-03-15; First posted 2011-11-22 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Respiratory Disorders
Keywords: Acute Lung Injury (ALI); Acute Respiratory Distress Syndrome (ARDS)
MeSH Terms: conditions — Respiration Disorders; Acute Lung Injury; Respiratory Distress Syndrome | interventions — GSK1995057

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK1995057 (Experimental): Single intravenous dose
  Interventions: Drug: GSK1995057 single dose
- Placebo (Placebo Comparator): Single intravenous dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK1995057 single dose — Single intravenous dose
  Arms: GSK1995057
Drug: Placebo — Single intravenous dose
  Arms: Placebo

SUMMARY:
The main purpose of the study is to see how safe GSK1995057 is and how well it is tolerated after dosing. The study will also investigate how GSK1995057 is taken up, metabolised (chemically broken down), distributed through the body and excreted, and what some of the effects of the study drug are.

DETAILED DESCRIPTION:
This study will be the first investigation of GSK1995057 in humans and is primarily designed to investigate safety and tolerability of single and repeat intravenously infused doses. The study will enrol healthy male subjects and healthy female subjects of non-child bearing potential and will also investigate immunogenicity, GSK1995057 distribution (pharmacokinetics), and potential impact on indicators of host immunity and normal immunological function. Safety, tolerability, immunogenicity, pharmacokinetic and pharmacodynamic data from this trial may facilitate further clinical investigations in healthy subjects dosed with GSK1995057 via the inhaled route, and ultimately clinical trials in patients with acute lung injury.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician.
* Male or female between 18 and 55 years of age inclusive
* A female subject is eligible to participate if she is of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation, hysterectomy or bilateral oophorectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea and elevated FSH as per the local laboratory guidelines.
* Normal creatinine clearance values at screening
* Male subjects must agree to use one of the study specific contraception methods
* Body weight ≥ 50 kg and BMI within the range 19 - 29.9 kg/m2 (inclusive).
* Normal lung function at screening.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Available to complete all study assessments.
* Able to read, comprehend and write English at a sufficient level to complete study elated materials.

Exclusion Criteria:

* A history of Hepatitis B, Hepatitis C or HIV infection and/or a positive pre-study HIV, Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities. (With the exception of known Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* Evidence of previous or active mycobacterium tuberculosis complex infection
* Recent history of and/or a positive test for Toxoplasma consistent with active oxoplasmosis infection.
* A positive test for influenza A/B taken within 7 days before dosing.
* Current evidence or history of an influenza-like illness.
* Corrected QT interval (QTcF) >450msec from ECG readings.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol and the following can be used as a guide: a half-pint (~240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.
* The subject is unwilling to abstain from alcohol consumption from 24 hr prior to dosing until discharge from the clinic, and for 24 hr prior to all other out-patient clinic visits.
* Subjects with a smoking history of >10 cigarettes per day in the last 3 months.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 90 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer) or exposure to more than four new chemical or biological entities within 12 months prior to the first dosing day.
* Subjects having received any type of vaccination within 3 weeks of the anticipated dosing start or are expected to be vaccinated within 3 weeks after the last dose.
* Current evidence of ongoing or acute infection, history of repeated or chronic significant infections or history of serious infection within three months of dosing.
* Subjects who have asthma or a history of asthma, COPD, other respiratory conditions or recurrent infections (a subject who suffered from childhood asthma but not as an adult may be included provided they fulfil other entry criteria).
* Subjects who have a known history of migraine headaches or are frequently suffering from other types of headaches which require medication (frequent defined as more than one headache in a fortnight).
* Use of prescription or non-prescription drugs (except simple analgesics), including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and sponsors Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy including severe allergic reaction, angio-edema or anaphylaxis that, in the opinion of the investigator or sponsors Medical Monitor, contraindicates their participation.
* History of malignancy, except for adequately treated non-invasive cancer of the skin (basal or squamous cell) or cervical carcinoma in situ (>2 yrs prior to dosing).
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 3 month or 90 day period.
* Subject is unable to refrain from travelling to countries with a high prevalence of TB or other areas of prevalent infectious disease as judged by the investigator or the sponsors medical monitor from the start of screening until the final follow-up visit.
* Subject is mentally or legally incapacitated.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2011-03-08 (Actual); Primary Completion 2012-06-17 (Actual); Study Completion 2012-06-17 (Actual)

PRIMARY OUTCOMES:
Occurance of adverse events. | From start of screening until 84 days after completion of single dose (Part A subjects) or first dose (Part B subjects).
  Number and type of adverse events recorded during study.
Change from baseline in blood pressure. | From start of screening until 28 days after completion of single or repeat dosing.
  Systolic and diastolic blood pressure values before and after dosing completion.
Change from baseline in heart rate. | From start of screening until 28 days after completion of single or repeat dosing.
  Heart rate before and after dosing completion.
Change from baseline in respiration rate. | From start of screening until 28 days after completion of single or repeat dosing.
  Respiration rate before and after dosing completion.
Change from baseline in body temperature. | From start of screening until 28 days after completion of single or repeat dosing.
  Body temperature before and after dosing completion.
Change from baseline in heart function. | For 24hrs during screening, then for 1 hour before dosing to 24 hours after dosing starts (in Part A subjects only, except for cohort 7).
  Holter recording.
Change from baseline in heart function | From 1 hour before dosing to 12 hours after dosing starts for each dose.
  Lead II cardiac telemetry.
Change from baseline in heart function. | From start of screening until 28 days after completion of single or repeat dosing.
  12-lead ECG recording.
Change from baseline in lung function. | From start of screening until 28 days after completion of single or repeat dosing.
  FEV1 and FVC measurements.
Change from baseline in laboratory safety data. | From start of screening until 28 days after completion of single or repeat dosing.
  Clinical chemistry, haematology and routine urinalysis.

SECONDARY OUTCOMES:
Plasma pharmacokinetics of GSK1995057 | From the first day of dosing until 48 hours after the completion of dosing.
  Levels of GSK1995057 in blood samples.
Urine pharmacokinetics of GSK1995057 | From 1 hour before the only dose until 48 hours after the dose.
  Levels of GSK1995057 in urine samples from cohort 6 subjects only.
Bronchoalveolar lavage fluid (BALF) (saline flushed into and then collected from a lung) pharmacokinetics. | At 2 hrs after the completion of the only dose.
  Levels of GSK1995057 in BALF from cohort 7 subjects only.
Effect of GSK1995057 on host immunity and immunological function | From the day before dosing starts to 28 days after dosing completion.
  Levels of pharmacodynamic and immune function biomarkers in blood samples.
Effects of GSK1995057 on host immunity and immunological function | At 2 hrs after the completion of the only dose.
  Levels of pharmacodynamic and immune function biomarkers in BALF from cohort 7 subjects only.
Immunogenic effect of GSK1995057 | From the start of screening (cohorts 1-4 only) or from the day before the start of dosing until 84 days after the completion of single or repeat dosing.
  Levels of anti-GSK1995057 antibodies in blood samples

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Harrow, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 110951 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/110951?search=study&search_terms=110951#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 110951 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110951 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110951 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110951 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 110951 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110951 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110951 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register